CLINICAL TRIAL: NCT03746054
Title: Phase III Study, Randomized, Multicenter, Evaluating the Efficacy of a Cardiovascular Active Prevention Vs Usual Clinical Practice, on the Morbi-mortality Decrease in Chronic Myeloid Leukemia Patients Treated with Tyrosine Kinase Inhibitor
Brief Title: Evaluation of a Cardiovascular Active Prevention in Chronic Myeloid Leukemia on the Cardiovascular Morbi-mortality
Acronym: PALERMO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inclusions stopped on 25MAR2022 due to lack of inclusion Last follow-up on 16APR2024
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC-K-2017
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: Blood; Chronic Myeloid Leukemia; Vascular medicine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active prevention (Experimental): optimal medical treatment
  Interventions: Combination Product: Optimal medical treatment
- usual clinical practice (Sham Comparator): usual clinical practice in each center
  Interventions: Combination Product: usual clinical practice

INTERVENTIONS:
Combination Product: Optimal medical treatment — Life style modifications, Monitoring of the risk factors and Optimal medical treatment Lipid-lowering treatment, anti-platelet treatment and ACEi or AT2 antagonists treatment for a total duration of 24 months
  Arms: active prevention
Combination Product: usual clinical practice — usual clinical practice in each center
  Arms: usual clinical practice

SUMMARY:
According to the French National Cancer Institute, 35 000 new hematologic cancers are observed in France representing 10% of the new cancers. Chronic Myeloid Leukemia (CML) is a cancer involving the bone marrow and blood cells, the median age at diagnosis is 53 years in the Western world. The prognosis is worse than many other cancers with net survival at 5 years of 26%.

Since the approval of imatinib, additional tyrosine kinase inhibitors (TKIs) have been approved by the European Medicine Agency, including the second-generation TKIs nilotinib, dasatinib, and bosutinib and the third-generation TKI ponatinib. Despite their effect on the evolution of CML, there is increasing of cardiovascular toxicities which can impact patient morbidity and mortality. The majority of the cardiovascular toxicities are associated with the second- and third-generation TKIs. Nilotinib and ponatinib cardiovascular toxicity including arterial and venous thromboembolism has decrease the benefit/risk ratio, 10% of patients treated with nilotinib 300 mg twice daily and 15.9% treated with 400 mg twice daily experienced a vascular complication including myocardial infarction /ischemic heart disease, cerebrovascular accidents, or peripheral arterial disease. Regarding ponatinib, serious arterial occlusive adverse reactions occurred in 19% of patients.

In an attempt to reduce major adverse cardiovascular events MACE due to nilotinib and ponatinib, currently, then approach is driven by usual clinical practice without any robust published evidence. The investigators aim to perform a national clinical trial, multicenter, prospective, randomized, with two parallel comparative arms: experimental group with cardiovascular active prevention vs non active cardiovascular active prevention based on usual clinical practice. Our hypothesis is that active prevention of cardiovascular toxicities with optimal medical treatment improves the benefit-risk ratio in CML patients. The primary objective is Event Free Survival (EFS) at month 24.

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed.

The efficacity of the cardiovascular active prevention will be studied by comparing the rate of Event free Survival between patients in the Experimental Arm Versus usual Clinical practices

The duration of participation for a subject is equal to 2 years

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* CML "Philadelphia chromosome" in chronic phase treated with nilotinib or ponatinib for, in first or second line
* Written informed consent must be obtained prior to protocol-specific procedures
* Affiliation to a social security category

Exclusion Criteria:

* Revascularization already decided and scheduled
* Life threatening disease
* Recent history of myocardial infarction or stroke
* Unstable angina
* Hypotension (Blood pressure < 90/50mmHg)
* Pregnancy and lactation
* Women of childbearing potential not using appropriate contraceptive measures
* Contraindication for statin
* Contraindication for aspirin
* Contraindication for ACEi or AT2 antagonists treatment
* Known hypersensitivity to rosuvastatin or fluvastatin, other ingredients in the product
* Known hypersensitivity to aspirin, other ingredients in the product, other salicylates or non-steroidal anti-inflammatory drugs
* Known hypersensitivity to ACEi or AT2 antagonists treatment, other ingredients in the product
* Hereditary or idiopathic angioedema ; or history of angioedema
* Hyperaldosteronism
* Active liver disease, or unexplained, persistent elevations in serum transaminases
* Severe renal impairment (creatinine clearance <30 ml/min)
* Myopathy
* Concomitant cyclosporine treatment
* History of gastrointestinal bleeding or perforation, related to previous NSAIDs therapy
* Severe heart failure
* Concurrent severe diseases which exclude the administration of therapy
* Patients under reinforced protection, deprived of liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social establishment for purposes other than research
* Absence of affiliation to a social security agency
* Inability to understand the instructions or objectives of the study
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Improvementof the Event Free Survival (EFS) rate in CML patients with an active and systematic prevention for cardiovascular risk. | 24 months
  The Event Free Survival (EFS) is based on the analysis of the time to an event occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: HENNI SAMIR, MD, PhD, Principal Investigator — Angers Teaching Hospital
Locations (1):
- CHU, Angers, France

IPD SHARING:
Plan to Share IPD: No